CLINICAL TRIAL: NCT02398305
Title: Shortening Compression Time of the Access Site After Cardiac Catheterisation Through the Radial Artery
Brief Title: Shortening Compression Time After Radial Access for Cardiac Catheterisation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, J.H.H. (Han) Deuling, MANP, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: METc2011-233
Record Dates: First submitted 2014-12-04; First posted 2015-03-25 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Cardiac Catheterisation
Keywords: Cardiac catheterisation; Radial access; Compression; Terumo TR Band; radial artery; diagnostic
MeSH Terms: conditions — Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TR Band accelerated (Active Comparator): Diminishing air pressure in the TR Band using accelerated protocol
  Interventions: Device: TR Band Quick
- TR band standard (Other): Diminishing air pressure in the TR band according to standard care
  Interventions: Device: TR Band standard

INTERVENTIONS:
Device: TR Band standard — Diminishing the air pressure in the TR Band following standard protocol
  Arms: TR band standard
Device: TR Band Quick — Diminishing the air pressure in the TR Band following a faster protocol
  Arms: TR Band accelerated

SUMMARY:
To obtain arterial access for a diagnostic cardiac catheterization or percutaneous coronary intervention (PCI) the cardiologist can choose between the femoral artery and the radial artery. In the University Medical Center Groningen the femoral artery is commonly used. After intervention the puncture site is closed with an arteriotomy closure device (ACD). Patients after radial access receive a pressure bandage at the puncture site, usually the Terumo (TR) wrist bandage.

The bedrest period for patients with an ACD is 1 hour after diagnostic cardiac catheterization and 2 hours after PCI. After the bedrest period patients are discharged 1 hour after diagnostic procedures or 4 hours after PCI. This to observe potential bleeding complications after the procedure. In patients with radial access, the TR bandage will be removed according to current protocol after 4 hours and additionally 1 hour observation is required. Several cardiologists have the intention to use the radial artery more frequent for cardiac catheterization or PCI. In a meta-analysis radial access is related to a 73% decrease in major bleeding complications compared to femoral access. Also there are no significant differences in MACE. Even so there are no differences in success percentage for cardiac catheterization or PCI and admission time is shorter for radial access (Am Heart J. 2009 Jan;157(1):132- 40). Admission time for diagnostic cardiac catheterization at the short-stay unit is in case of femoral access with an ACD approximately 2 hours. For patients after radial access post procedural admission time is approximately 5 hours. To guarantee patient throughput, uniformity of care and more efficient use of capacity of the short-stay unit, patients after radial access should not have a longer hospital admission time than patients after femoral access. Carrington et al. (J Interv Cardiol. 2009 Dec;22(6):571-5) have shown that it is safe to deflate the TR wrist band faster than four hours.

Objective of the study:

To describe the differences in safety, patient comfort and admission period after diagnostic cardiac catheterization through radial access, between the current protocol and the protocol of fast desufflation by Carrington et al.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic coronary angiogram
* Radial access
* 6 French sheath

Exclusion Criteria:

* Use of oral anticoagulants
* Percutaneous coronary intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2012-10; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Bleeding | 1 year
  Bleeding at puncture site after deflating pressure in TR band

SECONDARY OUTCOMES:
Swelling | 1 year
  Swelling at puncture site that is not caused by bleeding
Patient comfort | 1 year
  Patient comfort, measured on VAS
Time to discharge, after return on nursing unit | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pim van der Harst, MD PhD, Study Director — University Medical Center Groningen
Locations (1):
- University Medical Centre Groningen, Groningen, Provincie Groningen, Netherlands